CLINICAL TRIAL: NCT00251212
Title: Tailored Teen Alcohol and Violence Prevention in the ER
Brief Title: Tailored Teen Alcohol and Violence Prevention in the Emergency Room (ER)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Maureen A Walton, Associate Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AA-014889-01A1
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Violence; Alcohol Abuse
Keywords: Alcohol; Violence; Alcohol consumption; Alcohol, drinking
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Therapist delivered adapted motivational enhancement therapy and skills training
  Interventions: Behavioral: Adapted Motivational Interviewing & Skills Training
- 2 (Active Comparator): Computer delivered adapted motivational enhancement therapy and skills training
  Interventions: Behavioral: Adapted Motivational Interviewing & Skills Training
- 3 (No Intervention): 3: Control brochure

INTERVENTIONS:
Behavioral: Adapted Motivational Interviewing & Skills Training — Single session, 45 minute brief intervention during Emergency Department Visit
  Other Names: 1: Therapist delivered brief intervention; 2: Computer delivered brief intervention; 3: Control condition
  Arms: 1; 2

SUMMARY:
This study is designed to address both alcohol misuse and violence among adolescents ages 14-18 seeking care in an urban emergency department (ED). The study is a randomized controlled trial comparing the effectiveness of a combined Adapted Motivational Interviewing and Skills Training intervention, delivered either by a computer or by a counselor, and an informational handout control condition.

DETAILED DESCRIPTION:
This study will screen ~3000 adolescents in the ED (ages 14-18) over 30 months. Eligible adolescents will be asked to participate in the longitudinal study, stratified by age and gender and randomized to conditions (n=225/group): Computer Prevention Program, Counselor Prevention Program, or an informational handout control condition. Primary outcomes will be evaluated at 3, 6 and 12-months and include alcohol use/misuse, violent behaviors, illicit drug use, unintentional injury, delinquency, and weapon carriage. The proposed study integrates brief intervention strategies for alcohol misuse and violent behaviors using state-of-the-art technology to tailor the interventions to the specific risk factors of the adolescent. Tailored computerized programs use available technology to replace the need for clinical staff in the ED setting, where there is limited staff time to effect behavior change. This project will provide the critical first step toward the implementation of an integrated prevention program addressing overlapping risk factors that has the potential to be delivered to the millions of adolescents visiting urban Emergency Departments each year.

ELIGIBILITY:
Inclusion Criteria:

* adolescents (ages 14-18) presenting to the ED for a medical injury or illness (except exclusions as noted below)
* adolescents ability to provide informed assent/consent depending on age
* access to a parent or guardian to provide informed consent

Exclusion Criteria:

* adolescents who do not understand English
* prisoners
* adolescents classified by medical staff as "Level 1" trauma
* adolescents deemed unable to provide informed consent
* adolescents treated in the ED for suicide attempts
* adolescents triaged to the psychiatric ED

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3694 (Actual)
Dates: Start 2006-09; Primary Completion 2010-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome variables include alcohol misuse and violent behaviors. | 12-months

SECONDARY OUTCOMES:
Secondary outcome measures include illicit drug use, unintentional injury, delinquency and weapon carriage. | 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, PhD, MPH, Principal Investigator — University of Michigan

REFERENCES:
- [Background] Goldstein AL, Walton MA, Cunningham RM, Resko SM, Duan L. Correlates of gambling among youth in an inner-city emergency department. Psychol Addict Behav. 2009 Mar;23(1):113-21. doi: 10.1037/a0013912. PMID 19290695
- [Background] Walton MA, Cunningham RM, Goldstein AL, Chermack ST, Zimmerman MA, Bingham CR, Shope JT, Stanley R, Blow FC. Rates and correlates of violent behaviors among adolescents treated in an urban emergency department. J Adolesc Health. 2009 Jul;45(1):77-83. doi: 10.1016/j.jadohealth.2008.12.005. Epub 2009 Feb 20. PMID 19541253
- [Background] Whiteside LK, Walton MA, Stanley R, Resko SM, Chermack ST, Zimmerman MA, Cunningham RM. Dating aggression and risk behaviors among teenage girls seeking gynecologic care. Acad Emerg Med. 2009 Jul;16(7):632-8. doi: 10.1111/j.1553-2712.2009.00426.x. Epub 2009 Jun 9. PMID 19508314
- [Background] Resko SM, Walton MA, Bingham CR, Shope JT, Zimmerman M, Chermack ST, Blow FC, Cunningham RM. Alcohol availability and violence among inner-city adolescents: A multi-level analysis of the role of alcohol outlet density. Am J Community Psychol. 2010 Dec;46(3-4):253-62. doi: 10.1007/s10464-010-9353-6. PMID 20857328
- [Background] Cunningham RM, Resko SM, Harrison SR, Zimmerman M, Stanley R, Chermack ST, Walton MA. Screening adolescents in the emergency department for weapon carriage. Acad Emerg Med. 2010 Feb;17(2):168-76. doi: 10.1111/j.1553-2712.2009.00639.x. PMID 20370746
- [Background] Loh K, Walton MA, Harrison SR, Zimmerman M, Stanley R, Chermack ST, Cunningham RM. Prevalence and correlates of handgun access among adolescents seeking care in an urban emergency department. Accid Anal Prev. 2010 Mar;42(2):347-53. doi: 10.1016/j.aap.2009.11.012. Epub 2010 Jan 19. PMID 20159053
- [Background] Walton MA, Resko S, Whiteside L, Chermack ST, Zimmerman M, Cunningham RM. Sexual risk behaviors among teens at an urban emergency department: relationship with violent behaviors and substance use. J Adolesc Health. 2011 Mar;48(3):303-5. doi: 10.1016/j.jadohealth.2010.07.005. PMID 21338903
- [Background] Ranney ML, Whiteside L, Walton MA, Chermack ST, Zimmerman MA, Cunningham RM. Sex differences in characteristics of adolescents presenting to the emergency department with acute assault-related injury. Acad Emerg Med. 2011 Oct;18(10):1027-35. doi: 10.1111/j.1553-2712.2011.01165.x. PMID 21996067
- [Background] Resko SM, Walton MA, Chermack ST, Blow FC, Cunningham RM. Therapist competence and treatment adherence for a brief intervention addressing alcohol and violence among adolescents. J Subst Abuse Treat. 2012 Jun;42(4):429-37. doi: 10.1016/j.jsat.2011.09.006. Epub 2011 Nov 25. PMID 22119182
- [Background] Whiteside LK, Ranney ML, Chermack ST, Zimmerman MA, Cunningham RM, Walton MA. The overlap of youth violence among aggressive adolescents with past-year alcohol use-A latent class analysis: aggression and victimization in peer and dating violence in an inner city emergency department sample. J Stud Alcohol Drugs. 2013 Jan;74(1):125-35. doi: 10.15288/jsad.2013.74.125. PMID 23200158
- [Result] Cunningham RM, Walton MA, Goldstein A, Chermack ST, Shope JT, Bingham CR, Zimmerman MA, Blow FC. Three-month follow-up of brief computerized and therapist interventions for alcohol and violence among teens. Acad Emerg Med. 2009 Nov;16(11):1193-207. doi: 10.1111/j.1553-2712.2009.00513.x. PMID 20053240
- [Result] Walton MA, Chermack ST, Shope JT, Bingham CR, Zimmerman MA, Blow FC, Cunningham RM. Effects of a brief intervention for reducing violence and alcohol misuse among adolescents: a randomized controlled trial. JAMA. 2010 Aug 4;304(5):527-35. doi: 10.1001/jama.2010.1066. PMID 20682932
- [Result] Cunningham RM, Chermack ST, Zimmerman MA, Shope JT, Bingham CR, Blow FC, Walton MA. Brief motivational interviewing intervention for peer violence and alcohol use in teens: one-year follow-up. Pediatrics. 2012 Jun;129(6):1083-90. doi: 10.1542/peds.2011-3419. Epub 2012 May 21. PMID 22614776
- [Result] Cunningham RM, Whiteside LK, Chermack ST, Zimmerman MA, Shope JT, Bingham CR, Blow FC, Walton MA. Dating violence: outcomes following a brief motivational interviewing intervention among at-risk adolescents in an urban emergency department. Acad Emerg Med. 2013 Jun;20(6):562-9. doi: 10.1111/acem.12151. PMID 23758302
- [Derived] Stoddard SA, Whiteside L, Zimmerman MA, Cunningham RM, Chermack ST, Walton MA. The relationship between cumulative risk and promotive factors and violent behavior among urban adolescents. Am J Community Psychol. 2013 Mar;51(1-2):57-65. doi: 10.1007/s10464-012-9541-7. PMID 22744013